CLINICAL TRIAL: NCT05877326
Title: Anaesthetic Depth and Short Term Delirium Post Cardiac Surgery Intervention
Acronym: BISCAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Cardiologique du Nord (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A02200-43
Record Dates: First submitted 2023-05-02; First posted 2023-05-26 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Post-operative Delirium; Anaesthetic Depth
MeSH Terms: conditions — Emergence Delirium | interventions — Anesthesia, General; Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Multicenter, controlled, randomized, two parallel-arm trial:
  Perioperative anesthesia with a BIS target of 35 Perioperative anesthesia with a 55% BIS target
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative anesthesia with a BIS target of 35 (Active Comparator): Anesthesia with a BIS target of 35
  Interventions: Drug: General anesthesia with propofol or sevoflurane; Behavioral: CAM-ICU (Confusion Assesment Method ICU) at day 3 post-operative
- Perioperative anesthesia with a BIS target of 55 (Active Comparator): Anesthesia with a BIS target of 55
  Interventions: Drug: General anesthesia with propofol or sevoflurane; Behavioral: CAM-ICU (Confusion Assesment Method ICU) at day 3 post-operative

INTERVENTIONS:
Drug: General anesthesia with propofol or sevoflurane — General anesthesia
  Other Names: General anesthesia with 35 BIS target or 55 BIS target
Behavioral: CAM-ICU (Confusion Assesment Method ICU) at day 3 post-operative — The presence of mental confusion will be determined by CAM-ICU at J3 post intervention.

SUMMARY:
Postoperative delirium (POD) is a critical complication of major surgery and affects up to 70% of surgical patients over the age of 60 years.

The additional healthcare costs associated with delirium exceed €50,000 per patient per year due to prolonged hospital stay, increased risk of long-term care or institutionalization, and the risk of developing dementia or cognitive impairment . Therefore, prevention of POD is a major goal in the perioperative setting.

The investigator proposes this randomized study to evaluate the interest of a reduced anesthetic depth to prevent short-term cognitive disorders after cardiac surgery in elderly subjects.

Method: Patients over 75 years old scheduled to undergo one of the cardiac surgeries of interest (valvular, coronary bypass, aortic or combined surgery) will be randomized to 2 paralell arms :

* Perioperative anesthesia with a BIS (Bispectral index) target of 35
* Perioperative anesthesia with a BIS(Bispectral index) target of 55

The presence of mental confusion will be determined by CAM-ICU ( Confusion Assessment Method for the ICU ) at day 3 post procedure.

Ancillary study: To assess cognitive status at inclusion, discharge and third post operative month using the MOCA(Montreal Cognitive Assessment ).

Conclusion:The hypothesis of this study is that a lower depth of anesthesia will reduce post operative delirium in the first three days in patients older than 75 years who are planned for valvular, coronary artery bypass, aortic or combined cardiac surgery .

DETAILED DESCRIPTION:
Multicenter, controlled, randomized trial with two parallel arms (Perioperative anesthesia with a BIS target of 35 / Perioperative anesthesia with a BIS target of 55).

Randomization will be stratified by center, type of surgery (valve vs coronary artery bypass surgery vs aortic surgery vs combined surgery), patient age (75-80 vs 81-85), Euroscore 2 score at inclusion (predicted mortality risk ≥ vs < to 30%).

An ancillary study with MOCA score measurement at inclusion, discharge and 3 months after cardiac surgery will be realized.

Primary Objective:

To demonstrate the benefit of lower anesthesia on the prevalence of delirium during the first 3 days postoperatively in patients aged 75 years and older having cardiac surgery (valvular, coronary bypass, aortic or combined surgery).

Primary endpoint:

Presence of mental confusion will be determined by CAM-ICU at day 3 post surgery.

The CAM-ICU is considered POSITIVE (confusion present) if criteria 1 and 2 + 3 or 4 are met.

Secondary objectives:

To evaluate the effects of the intervention on ICU and hospital length of stay, delirium durations, mortality at month 3 , prevalence of POD during the stay, duration of mechanical ventilation, rate of reintubation,total amount of propofol, opioids and neuromuscular blockade (au lieu de curares) during anesthesia .

Secondary endpoints:

CAM ICU at times day 1, Day 2 , and Day 3 , daily doses of benzodiazepines, opiates, propofol, dexmedetomidine, and neuroleptics, days without mechanical ventilation, ICU and total lengths of stay, vital status (phone call) at Month 3, duration of delirium, total amount of propofol, opioids and neuromuscular blockade during anesthesia .

In order to demonstrate a minimum difference in the confounding rate (according to CAM-ICU) of 20 points (50% expected in the BIS 35 arm versus 30% in the BIS 55 arm) and with a two-sided first-species risk of 5% and a minimum power of 80%, 186 analyzable subjects (93 per arm) are required.

In order to take into account possible loss of sight, we propose to include in this study a total of 200 subjects (100 per arm).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 75 and 85 years, who signed an informed consent, undergoing elective valvular, coronary artery bypass, aortic or combined cardiac surgery
* Be affiliated to French Health Insurance

Exclusion Criteria:

* Refusal of consent -Patient unable to read, write or understand French
* Vulnerable patient according to article L1121-6 of the CSP,
* Patient of legal age under guardianship or curatorship or under legal protection,
* Patient unable to give personal consent according to article L.1121-8 of the CSP or adult protected by law,
* Patient having already participated in the present study

Ages: 75 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the benefit of reduced depth of anesthesia | Day 3 post intervention.
  The presence of mental confusion using CAM-ICU ( The Confusion Assessment Method for the Intensive Care Unit )

CONTACTS AND LOCATIONS:
Overall Officials: Ellouze Omar, MD, Principal Investigator — Centre Cardiologique du Nord
Locations (1):
- Centre cardiologique du nord, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No
The sponsor and the persons acting on its behalf will have access to the data. In addition, only the persons delegated by the investigating physician, health or research professionals, involved in the realization of the research and subject to professional secrecy, will have access to these coded data.

REFERENCES:
- [Derived] Ellouze O, Zogheib E, Abdelhafidh K, Lemaire A, Berger J, Charfeddine A, Bouzguenda H, Konstantinou M, Molinari N, Bonnet N, Geri G, Nappi F. Anaesthetic depth and short-term delirium after cardiac surgery intervention: the study protocol of the BISCAR multicentre randomised clinical trial. BMJ Open. 2025 Aug 28;15(8):e103105. doi: 10.1136/bmjopen-2025-103105. PMID 40876878